CLINICAL TRIAL: NCT00814008
Title: The Relationship Between Stage of Diabetic Retinopathy and Retinal Blood Flow in Patients With IDDM During Euglycemic Clamp
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Hans-Georg Eichler, MD, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OPHT-181298
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes Mellitus, Type 1; Insulin; Retina; Regional Blood Flow
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin; Glucose

INTERVENTIONS:
Drug: Insulin — Insulin Dosage form : intravenous infusion, infusion period 60 minutes Dosage: continuous dose of 0.5 mU/kg/min infused intravenously over 60 min; Insulin Lilly, Huminsulin, Lilly, Fegersheim, France
Drug: Glucose — Glucose:
  Dosage form : intravenous infusion, infusion period 60 minutes per dose level Dosage: at a rate to maintain blood glucose level at 100mg ; 20mg/100ml Glucose

SUMMARY:
Impaired retinal blood flow has been implicated in the pathogenesis of diabetic retinopathy. Patel et al. (1992) showed that retinal blood flow increases with the level of diabetic retinopathy. Grunwald et al. (1996) reported that patients with insulin dependent diabetes mellitus (IDDM) of relatively short duration have increased retinal blood flow, even before the onset of diabetic retinopathy. On the other hand the data of Bursell et al. (1996) indicate that IDDM patients have reduced retinal blood flow, when they have normal blood glucose levels, but this study may have considerable methodological limitations. Acute elevations of blood glucose levels, however, result in an increase in retinal blood flow (Grunwald et al. 1987, Bursell et al. 1996). Based on previous experimental data the investigators hypothesize that ocular blood flow is increased in early diabetes and reduced at later stages of the disease. Previous studies have demonstrated that metabolic conditions such as hyperglycemia influence outcome parameters and thereby might have confounded results regarding ocular blood flow in diabetic retinopathy. The investigators will therefore study patients with IDDM during euglycemic conditions.

ELIGIBILITY:
Inclusion Criteria:

Patients with IDDM:

* Age >= 19 years
* Best corrected visual acuity >= 0.8
* Ametropia < 6 dpt

Healthy control subjects:

* Age and sex matched to the subjects in the patients group
* Best corrected visual acuity >= 0.8
* Ametropia < 6 dpt

Exclusion Criteria:

Any of the following will exclude a diabetic patient from the study:

* Presence of intraocular pathology other than diabetic retinopathy (for example: cataract, glaucoma, ocular hypertension)
* Hypertension (Systolic blood pressure > 160 mm Hg or diastolic blood pressure > 90 mm Hg)
* Previous laser photocoagulation treatment
* Pregnancy (in women)

Any of the following will exclude a healthy subject from the study:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* Pregnancy (in women)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 1999-03; Primary Completion 2000-04 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
retinal blood flow after 1 hour of insulin clamp | 2 x 2 minutes

SECONDARY OUTCOMES:
Mean blood velocities in ophthalmic artery, posterior ciliary arteries and central retinal artery after 1 hour of insulin clamp | 2 x 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Georg Eichler, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria